CLINICAL TRIAL: NCT07267780
Title: The Contribution of Oncovascular Surgery in the Treatment of Gynecological Advanced Malignant Diseases: a Prospective and Retrospective Multicenter Study
Brief Title: Contribution of Oncovascular Surgery in the Treatment of Gynecological Advanced Malignant Diseases.
Status: Not yet recruiting | Type: Observational
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Other Study IDs: ONCOVASCULAR SURGERY
Record Dates: First submitted 2025-09-22; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Ovarian Carcinoma; Cervical Carcinoma; Endometrial Carcinoma; Vulvar Carcinoma; Uterine Sarcoma; Gynecologic Tumor
Keywords: Advanced or recurrent gynecologic tumor; Vascular infiltration
MeSH Terms: conditions — Ovarian Neoplasms; Uterine Cervical Neoplasms; Endometrial Neoplasms; Vulvar Neoplasms; Genital Neoplasms, Female

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective Arm (30 patients): Includes patients who underwent surgical treatment in the 8 years prior to the prospective study (January 1, 2017 - August 31, 2025).
- Prospective Arm (100 patients)

SUMMARY:
Multicenter ambispective observational study (prospective/retrospective)

DETAILED DESCRIPTION:
This multicenter ambispective observational study, including both a retrospective phase (patients treated surgically between January 1, 2017, and August 31, 2025) and a prospective phase, aims to evaluate the role of onco-vascular surgery in the treatment of advanced and recurrent gynecologic cancers. Onco-vascular surgery involves the simultaneous resection and reconstruction of major blood vessels when the tumor infiltrates or adheres firmly to them, and its benefits have been demonstrated in other malignancies such as hepatobiliary-pancreatic cancers and retroperitoneal soft tissue sarcomas. In the context of gynecologic oncology, this surgical approach is an emerging field with the potential to increase the rate of complete (R0) resection without increasing morbidity or mortality. However, data on the frequency, safety, and oncologic outcomes of vascular surgery in gynecologic oncology remain limited.

The study collects data on patient demographics, tumor characteristics, surgical details, postoperative complications, adjuvant therapies, oncologic outcomes, and quality of life (EORTC QLQ-C30).

Primary Objective: To describe overall survival in patients with advanced or recurrent gynecologic cancers undergoing onco-vascular surgery. Additionally, survival outcomes-including overall survival and 5-year progression-free survival-will be assessed for each patient subgroup, stratified by gynecologic cancer type and disease status (initial diagnosis vs. recurrence).

ELIGIBILITY:
Inclusion Criteria:

- Retrospective Arm:

1. Diagnosis of advanced or recurrent gynecologic cancer with vascular involvement requiring resection and/or reconstruction of major blood vessels, including:

   * Ovarian carcinoma
   * Cervical carcinoma
   * Endometrial carcinoma
   * Vulvar carcinoma
   * Uterine or other types of sarcomas with vascular involvement
2. Documented major vascular invasion, confirmed by preoperative imaging or intraoperative description.
3. Patients who underwent onco-vascular surgery for advanced or recurrent gynecologic cancers between January 1, 2017, and August 31, 2025.
4. Data Protection Impact Assessment (DPIA) approved for the management of retrospective data. (Deceased or untraceable patients will also be included to avoid selection bias, in accordance with Article 110 bis, paragraph 4 of the Italian Privacy Code. A DPIA will be produced and published on the Sponsor's website before study initiation, and patients who explicitly objected before death will not be included.)

Prospective Arm:

1. Age ≥18 years
2. Patients eligible for onco-vascular surgery for advanced or recurrent gynecologic cancers with vascular involvement, including:

   * Ovarian carcinoma
   * Cervical carcinoma
   * Endometrial carcinoma
   * Vulvar carcinoma
   * Uterine or other types of sarcomas
3. Documented major vascular invasion, confirmed by preoperative imaging or intraoperative description.
4. Signed informed consent.

Exclusion Criteria:

1. Patients younger than 18 years of age
2. Patients with early-stage gynecologic cancers not eligible for onco-vascular surgery
3. Patients undergoing vascular resection due to accidental injury of blood vessels not directly related to tumor infiltration.
4. Patients who have previously undergone vascular surgery for reasons unrelated to the study, to avoid data overlap.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population of the study consists of patients with advanced or recurrent gynecologic cancers involving major blood vessels by continuity or contiguity, who undergo en bloc tumor resection with simultaneous vascular resection and reconstruction during surgery for disease management.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2030-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | 5 years from the date of surgery
  Overall Survival (OS) at 5 years post-surgery, defined as the time from the surgical intervention to death from any cause. For patients who are still alive, OS will be censored at the date of the last follow-up.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | 5 years from the date of surgery
  Progression-Free Survival (PFS) at 5 years post-surgery Defined as the time from surgery to the first detection of recurrence or death, whichever occurs first. For patients without events, PFS will be censored at the date of the last follow-u
Frequency of early postoperative complications | 30 days post-surgery
  Complications will be classified according to the Clavien-Dindo system
Frequency of late postoperative complications | 180 days post-surgery
  Complications will be classified according to the Clavien-Dindo system.
Quality of Life assessment using the EORTC QLQ-C30 questionnaire | Baseline (30 days pre-surgery) and 1 month, 3 months, 6 months ans 12 months post-surgery
  Questionnaire administration
Number of days of postoperative hospital stay | From the date of surgery until post-operative hospital discharge(assessed up to 30 days after surgery)

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Istituto Nazionale Tumori IRCCS Fondazione G. Pascale, Napoli, Campania
  - A.R.N.A.S. Ospedali Civico Di Cristina Benfratell, Palermo, Italy